CLINICAL TRIAL: NCT06809179
Title: A Phase 2, Three-arm, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy, Safety, and Tolerability of a Repeat Dose of Fasedienol (PH94B) Nasal Spray for the Acute Treatment of Anxiety Induced by a Public Speaking Challenge in Adult Subjects With Social Anxiety Disorder, With an Open-Label Extension
Brief Title: A Clinical Trial to Assess the Efficacy, Safety, and Tolerability of a Repeat Dose of Fasedienol Nasal Spray for the Acute Treatment of Anxiety in Adults With Social Anxiety Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: VistaGen Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PH94B-CL036
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Social Anxiety Disorder
Keywords: Fasedienol; PH94B; social anxiety disorder; social anxiety; SAD; pherine; pherine nasal spray; acute treatment; anxiolytic; mental health; performance anxiety; anxiety nasal spray; anxiety treatment; public speaking anxiety; social phobia; phobic disorders; mental disorder; speech task
MeSH Terms: conditions — Phobia, Social; Psychological Well-Being; Phobic Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Fasedienol Nasal Spray (single dose) (Experimental): Twenty minutes prior to the PSC, subjects will receive one dose of Fasedienol Nasal Spray followed by one dose of Placebo Nasal Spray, separated by 10-minutes in between the two doses.
  Interventions: Drug: Fasedienol Nasal Spray - Placebo Nasal Spray
- Fasedienol Nasal Spray (repeat dose) (Experimental): Twenty minutes prior to the PSC, subjects will receive one dose of Fasedienol Nasal Spray followed by a second dose of Fasedienol Nasal Spray, separated by 10-minutes in between the two doses.
  Interventions: Drug: Fasedienol Nasal Spray - Fasedienol Nasal Spray
- Placebo Nasal Spray (Experimental): Twenty minutes prior to the PSC, subjects will receive one dose of Placebo Nasal Spray followed by a second dose of Placebo Nasal Spray, separated by 10-minutes between the two doses.
  Interventions: Drug: Placebo Nasal Spray - Placebo Nasal Spray

INTERVENTIONS:
Drug: Fasedienol Nasal Spray - Placebo Nasal Spray — Twenty minutes prior to the PSC, subjects will receive one dose of Fasedienol Nasal Spray followed by one dose of Placebo Nasal Spray, separated by 10-minutes in between the two doses.
  Arms: Fasedienol Nasal Spray (single dose)
Drug: Fasedienol Nasal Spray - Fasedienol Nasal Spray — Twenty minutes prior to the PSC, subjects will receive one dose of Fasedienol Nasal Spray followed by a second dose of Fasedienol Nasal Spray, separated by 10-minutes in between the two doses.
  Arms: Fasedienol Nasal Spray (repeat dose)
Drug: Placebo Nasal Spray - Placebo Nasal Spray — Twenty minutes prior to the PSC, subjects will receive one dose of Placebo Nasal Spray followed by a second dose of Placebo Nasal Spray, separated by 10-minutes between the two doses.
  Arms: Placebo Nasal Spray

SUMMARY:
This U.S. multicenter, double-blind, placebo-controlled Phase 2 clinical trial is designed to evaluate the efficacy, safety, and tolerability of a repeat intranasal (i.n.) dose of Fasedienol Nasal Spray (fasedienol) (3.2 µg) to relieve symptoms of acute anxiety in adult subjects ages 18 through 65 with Social Anxiety Disorder induced by a public speaking challenge (PSC) in a clinical setting. In addition, safety and tolerability of i.n. administration of 3.2 µg of fasedienol, as-needed, up to 6 times per day for up to 12 months, will be assessed in those subjects who complete PH94B-CL036 and choose to enter the distinct open-label extension phase of the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent provided prior to conducting any study-specific assessment.
* Male and female adults, 18 through 65 years of age, inclusive.
* Current diagnosis of SAD as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, and confirmed by the Mini-International Neuropsychiatric Interview (MINI).
* Clinician-rated Liebowitz Social Anxiety Score (LSAS) total score ≥70 at Screening (Visit 1).
* Clinician-rated Hamilton Depression Rating Scale (HAM-D) (17-items) total score <16.
* Female subjects of childbearing potential must be able to commit to the consistent and correct use of an effective method of birth control throughout the study
* Subjects must have normal olfactory function

Exclusion Criteria:

* Any history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, psychosis, anorexia or bulimia, premenstrual dysphoric disorder, autism spectrum disorder, or obsessive-compulsive disorder.
* Any other current principal or personality disorder (previously known as Axis I or Axis II disorders), except for specific phobias or generalized anxiety disorder, provided that these are not the primary diagnosis.
* Subjects who meet criteria for moderate or severe alcohol use disorder within the 1 year prior to study entry, or any use of illicit substances or tetrahydrocannabinol ("THC") within 2 months prior to study entry.
* In the opinion of the investigator, the subject has a significant risk for suicidal behavior during the course of their participation in the study, or the subject is considered to be an imminent danger to themself or others.
* Clinically significant nasal pathology or history of significant nasal trauma, nasal surgery, total anosmia, or nasal septum perforation that may have damaged the nasal chemosensory epithelium.
* Two or more documented failed adequate treatment trials with a registered medication approved for SAD.
* Currently receiving cognitive-behavioral therapy (CBT), exposure therapy, or acceptance and commitment therapy.
* Subjects taking psychotropic medications within 30 days before Visit 2.
* Use of any over-the-counter product, prescription product, off-label treatment, cannabidiol ("CBD"), or herbal preparation for treatment of the symptoms of anxiety or social anxiety within 30 days before Visit 2.
* Prior participation in a clinical trial involving fasedienol.
* Participation in any other clinical trial within the last 30 days or during the course of the current trial.
* Subjects with a positive urine drug screen.
* Women who have a positive urine pregnancy test.
* Women who are currently breastfeeding are not eligible unless they are willing to stop breastfeeding for the duration of the study.
* Subjects who have tested positive and/or have exhibited symptoms consistent with SARS-CoV-2 infection during the 4 weeks prior to Screening (Visit 1).
* Any clinically significant medical history or findings as determined by the Investigator that could interfere with the objectives of the study or put the participant at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 7 days (Visit 2 to Visit 3)
  The SUDS is a patient self-rated acute measurement scale that is scored in the range of 0 to 100 (operationalized for participants in this study as 0=totally relaxed or no anxiety at all and 100=highest distress or anxiety ever felt.

SECONDARY OUTCOMES:
Global Impression Scale of Improvement (CGI-I) | 7 days (Visit 2 to Visit 3)
  The CGI-I scale is a clinician-rated scale to assess illness improvement. The CGI-I scale includes one item being scored from 1 (best outcome) to 7 (worst outcome) with 4 being no change.
Patient Global Impression of Change (PGI-C) | 7 days (Visit 2 to Visit 3)
  The PGI-C is a patient self-rated scale to assess improvement. The PGI-C includes 7 items being scored from 1 (best outcome) to 7 (worst outcome) with 4 being no change.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Vistagen Clinical Site, Sherman Oaks, California
  - Vistagen Clinical Site, Walnut Creek, California
  - Vistagen Clinical Site, Largo, Florida
  - Vistagen Clinical Site, Saint Charles, Missouri
  - Vistagen Clinical Site, Toms River, New Jersey
  - Vistagen Clinical Site, Cary, North Carolina
  - Vistagen Clinical Site, Cleveland, Ohio
  - Vistagen Clinical Site, Plymouth Meeting, Pennsylvania
  - Vistagen Clinical Site, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.socialanxietytrials.com